CLINICAL TRIAL: NCT05633771
Title: A Multicenter, International, Prospective, Non-interventional, Observational Study, to Assess Treatment Retention of an Adalimumab Biosimilar (Hyrimoz®) in IBD Patients in Real Life Setting
Brief Title: Observational Study, to Assess Treatment Retention of an Adalimumab Biosimilar (Hyrimoz®) in IBD Patients in Real Life Setting
Acronym: HYRISS
Status: Active, not recruiting | Type: Observational
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Other Study IDs: CGP2017IC01
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; IBD; NIS; HYRISS; adalimumab; Hyrimoz
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — adalimumab biosimilar HS016

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hyrimoz: Patients prescribed with Hyrimoz
  Interventions: Other: Hyrimoz

INTERVENTIONS:
Other: Hyrimoz — There is no treatment allocation. Patients administered Hyrimoz by prescription that have started as routine medical treatment will be enrolled.
  Other Names: adalimumab biosimilar

SUMMARY:
An international, multicenter, non-interventional, prospective, post-authorization, descriptive, non-PASS, study.

DETAILED DESCRIPTION:
The main purpose of this non-interventional study is to assess patient retention with Hyrimoz® treatment up to 6 months after treatment initiation in Inflammatory Bowel Disease (IBD) patients.

Primary data will be collected at each data collection time point (visits will be according to local clinical practice). Data will be collected based on the information reported in the medical records. This study does not impose a therapy protocol, procedure or change in routine medical practice. Apart from self-administered questionnaires, no additional examinations or assessments are required, consequently there are no additional medical risks for the patients. The total duration of the study will be 36 months (3 years). The recruitment period will be for 2 years with individual patient follow-up for up to 1 year.

It is expected that patients will visit their physicians at regular intervals depending on local specific clinical practices. Four time points for data collection will be defined:

* T0 (patient inclusion in the study and Baseline characteristics).
* T1 (3-month follow-up ± 1 month).
* T2 (6-month follow-up and primary criteria -2/+3 months).
* T3 (12-month follow-up -3/+2 months).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria at Baseline:

* Patients initiating Hyrimoz® treatment.
* Patients with a confirmed diagnosis (following local recommendations) of one of these indications: CD or UC.
* Patients ≥ 18 years of age.
* Patient in whom the decision to initiate Hyrimoz® (naïve population) or to switch (switch population) from reference adalimumab to Hyrimoz® was accorded with his physician before the proposal to participate in the study.
* Patients meeting one of the following criteria:

  * Referred to as "switched patients": Patients treated continuously with adalimumab (other than Hyrimoz®) for at least 6 months, with an indication for continuing treatment with adalimumab at any therapeutic dose (physician's decision) and who have controlled stable disease for at least 3 months before study enrollment (according to the physician's criteria).
  * Referred to as "biologic-naive patients": Patients who had an inadequate response or contraindications to conventional therapy with no exposure to any biological medicine and targeted therapies and started Hyrimoz® as a first-line biologic therapy according to the summary of product characteristics (SmPC).
* Patients able to complete and understand the self-administered questionnaires.
* Patients who have been informed and have provided a signed written consent as per local regulations prior to participation in the study

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Patients enrolled in an ongoing interventional study.
* Patients with any contraindications to Hyrimoz® according to the SmPC.
* Patients at imminent risk of scheduled intestinal surgery (stenosis, strictures, internal fistula).
* Use of any investigational drug in last 6 months prior to enrollment.
* Patient received any biological medicine or targeted therapy, in case of " biologic-naive patient ",
* Patient received adalimumab for less than 6 months or have controlled disease for less than 3 months, in case of "switched patient".

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom the investigator has decided to initiate treatment with Hyrimoz® in accordance with the approved SmPC and local clinical practice, will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who remain on Hyrimoz® at 6 months after treatment initiation | Up to 6 months
  Assess patient retention with Hyrimoz® treatment up to 6 months after treatment initiation

SECONDARY OUTCOMES:
Percentage of patients who discontinue Hyrimoz | 6 months, 12 months
  Percentage of patients who discontinue Hyrimoz® at T2 and T3 due to:
  * Lack of efficacy.
  * Intolerance/Adverse event(s) or special scenario.
  * Patient's decision
  * Nocebo effect
  * Other reasons.
Percentage of patients with high level of treatment satisfaction using TSQM-9 questionnaire | 3 months, 6 months, 12 months
  To assess patients' treatment satisfaction (based on 9-item Treatment Satisfaction Questionnaire for Medication [TSQM 9], the percentage of patients with high level of treatment satisfaction (score ≥ 39) will be collected.
  The TSQM-9 is declined with 9 questions about patient treatment satisfaction. Each answer gives a number of points depending of the question and the answer. The final score is the sum of points in each question. This questionnaire score from 9 to 59 points. In HYRISS study, we estimate that patient with < 39 pts in TSQM-9 are considered with a low satisfaction for the medication (satisfaction under 60%).
Percentage of patients with high level of treatment adherence using adapted CQR5 questionnaire | Baseline, 3 months, 6 months, 12 months
  To assess adherence/compliance to treatment (based on 5 item Compliance Questionnaire for Rheumatology [CQR5] adapted for gastroenterologist), percentage of patients with high level of treatment adherence (score ≥ 15) using adapted CQR5 questionnaire will be collected.
  The CQR5 is declined with 5 questions about patient compliance to the treatment. Each answer gives from 1 to 4 points depending of the answer. The final score is the sum of points in each question. This questionnaire score from 5 (very low compliance) to 20 points (very strong compliance).
Percentage of patients with the perception of a high level of disease activity using VAS scale | Baseline, 3 months, 6 months, 12 months
  To assess the patient's reported disease activity, percentage of patients with the perception of a high level (score ≥ 6) of disease activity will be collected using visual analog scale [VAS].
  This visual analogue scale (VAS) is an instrument designed to document the disease activity. Patients are asked to rate their disease activity on a visual analogue scale (VAS): How active has your disease been this week? From 0 (Not active at all) to 10 cm (Extremely active).
Percentage of patients with a good perception about biosimilars using VAS scale | Baseline
  To assess the patient's reported perception about biosimilars at the inclusion visit, percentage of patients with a good perception (score ≥ 6) about biosimilars using VAS scale will be measured.
  This visual analogue scale (VAS) is an instrument designed to document the perception of the patient about biosimilar. Patients are asked to rate their perception of biosimilar medicine on a visual analogue scale (VAS): Are you confident in using biosimilar? From 0 (I have no confidence at all) to 10 cm (I have a great confidence).
Percentage of patients in remission | Baseline, 3 months, 6 months, 12 months
  Remission defined as Harvey-Bradshaw Index [HBI] ≤ 4 [for Crohn's Disease] or partial Mayo score ≤ 1 [for Ulcerative Colitis]
Crohn's disease activity measurement: Harvey Bradshaw Index [HBI] | Up to 12 months
  Crohn's disease activity will be measured with HBI score. Score is interpreted:
  <4: Remission 4-7: Mild disease 8-16: Moderate disease >16: Severe disease
Ulcerative colitis activity measurement: partial Mayo calculation score | Up to 12 months
  Ulcerative colitis activity will be measured using partial Mayo calculation score. Score is interpreted: ≤ 1: Remission 2 - 4: Low activity disease 5 -6: Moderate disease 7 - 9: Severe disease
Pattern of Hyrimoz® utilization | Up to 12 months
  Pattern of Hyrimoz® utilization to be collected

CONTACTS AND LOCATIONS:
Locations (51):
- Belgium (13):
  - Sandoz Investigational Site Belgium, Aalst
  - Sandoz Investigational Site Belgium, Antwerp
  - Sandoz Investigational Site Belgium, Bonheiden
  - Sandoz Investigational Site Belgium, Brussels
  - Sandoz Investigational Site Belgium, Eeklo
  - Sandoz Investigational Site Belgium, Ghent
  - Sandoz Investigational Site Belgium, Herentals
  - Sandoz Investigational Site Belgium, Kortrijk
  - Sandoz Investigational Site Belgium, Liège
  - Sandoz Investigational Site Belgium, Namur
  - Sandoz Investigational Site Belgium, Seraing
  - Sandoz Investigational Site Belgium, Sint-Niklaas
  - Sandoz Investigational Site Belgium, Tongeren
- France (38):
  - Sandoz Investigational Site France, Amiens
  - Sandoz Investigational Site France, Auxerre
  - Sandoz Investigational Site France, Bayonne
  - Sandoz Investigational Site France, Beauvais
  - Sandoz Investigational Site France, Brest
  - Sandoz Investigational Site France, Caen
  - Sandoz Investigational Site France, Castelnau-le-Lez
  - Sandoz Investigational Site France, Clermont-Ferrand
  - Sandoz Investigational Site France, Clichy
  - Sandoz Investigational Site France, Cornebarrieu
  - Sandoz Investigational Site France, Créteil
  - Sandoz Investigational Site France, Gien
  - Sandoz Investigational Site France, Le Coudray
  - Sandoz Investigational Site France, Le Kremlin-Bicêtre
  - Sandoz Investigational Site France, Lille
  - Sandoz Investigational Site France, Lyon
  - Sandoz Investigational Site France, Marseille
  - Sandoz Investigational Site France, Montpellier
  - Sandoz Investigational Site France, Nancy
  - Sandoz Investigational Site France, Neuilly-sur-Seine
  - Sandoz Investigational Site France, Nice
  - Sandoz Investigational Site France, Nîmes
  - Sandoz Investigational Site France, Orléans
  - Sandoz Investigational Site France, Paris
  - Sandoz Investigational Site France, Pessac
  - Sandoz Investigational Site France, Pierre-Bénite
  - Sandoz Investigational Site France, Poitiers
  - Sandoz Investigational Site France, Pringy
  - Sandoz Investigational Site France, Reims
  - Sandoz Investigational Site France, Rennes
  - Sandoz Investigational Site France, Saint-Etienne
  - Sandoz Investigational Site France, Saint-Nazaire
  - Sandoz Investigational Site France, Sarrebourg
  - Sandoz Investigational Site France, Toulouse
  - Sandoz Investigational Site France, Tours
  - Sandoz Investigational Site France, Troyes
  - Sandoz Investigational Site France, Vandœuvre-lès-Nancy
  - Sandoz Investigational Site France, Vénissieux

IPD SHARING:
Plan to Share IPD: No